CLINICAL TRIAL: NCT02692287
Title: The Postpartum Haemorrhage (PPH) Butterfly Work Package 3, Phase I in Vivo Testing
Brief Title: The Postpartum Haemorrhage (PPH) Butterfly Work Package 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Weeks MD MRCOG (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Andrew Weeks MD MRCOG, Professor of International Maternal Health, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: V.2.4
Record Dates: First submitted 2016-02-12; First posted 2016-02-26 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Postpartum Haemorrhage (PPH)
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: If the device is not of the correct size, then the device is changed and the recruitment process is repeated until the correct size is obtained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the PPH Butterfly (Other): The PPH Butterfly will be inserted into the vagina of a healthy postnatal woman
  Interventions: Device: The PPH Butterfly

INTERVENTIONS:
Device: The PPH Butterfly — The PPH Butterfly is a simple, low cost device that has been developed to facilitate less invasive compression of the uterus in a PPH

SUMMARY:
The Postpartum Haemorrhage (PPH) Butterfly is a simple, low-cost device which has been developed as a treatment method for PPH. It will be used to stop the bleeding through compression of the uterus of women having a PPH. It will be markedly easier to undertake than traditional bimanual compression, whilst also being significantly more acceptable to women themselves. Use of the PPH Butterfly will provide an alternative management option for PPH and in some cases should avoid the need for women to have to go to theatre for treatment. This research will allow the investigators to determine if they have the optimum size and shape of the device, that it will operate as intended when compressing the uterus, and to gauge its acceptability to participants and users. In phase I the investigators will recruit "healthy volunteers" i.e. women who have delivered their baby vaginally following Induction of labour (IOL) however these women will not be experiencing a PPH. The device is to be assessed purely on size, usability and acceptability not for diagnosis or as a treatment method. Following the delivery participants will be invited to have the PPH Butterfly inserted vaginally for an average of 2 minutes. It is through this that the investigators will assess the suitability of the device in its current design, when it is in practice. The clinician who operates the device will complete a Likert scale questionnaire along with some open questions following each administration. Participants will also answer a short questionnaire. .

DETAILED DESCRIPTION:
The study will involve 5-10 healthy women who deliver their baby vaginally following Induction of Labour (IOL). The women will be given a short leaflet regarding the study. During their time on the Induction of Labour (IOL) Suite, women will be seen by a member of the research team, the research will be discussed with them and they will receive a Participant Information Sheet if they desire. The woman will also be shown a short video regarding the Postpartum Haemorrhage (PPH)Butterfly which is specifically for members of the public. After a discussion of the research, women will be asked to indicate in writing whether they may consider participation, whether they do not want to participate, or whether they are undecided but are happy to be asked again. Only those women who are considering participation, or who are happy to be asked again will be approached post-delivery. All of the women can be approached up to 72 hours post-delivery and asked if they wish to participate. If a woman has a vaginal delivery, a member of the research team will then attend the Delivery Suite, maternity theatre (the woman may have had an instrumental delivery in theatre) or the postnatal ward once informed by the midwife caring for her. They will clarify with the woman if she wishes to participate. Assuming the woman wishes to participate, informed, signed consent will be sought at this point and the device will be used, with a speculum examination taking place before and after use of the device.

If the device is of an incorrect size, then the device size will be changed before repeating the process with 5-10 more women. In this way the final recruitment number may be more than 10 in total.

ELIGIBILITY:
Inclusion Criteria:

* Women who have a vaginal delivery following induction of labour and who are within 72 hours of delivery.

Exclusion Criteria:

* Women assessed antenatally to have learning difficulties that may have the potential to impair their decision making
* Women aged < 16 years of age
* Women who cannot read or understand the level of English used in the study documentation
* Women who've had a stillbirth (in this pregnancy)
* Women who have undergone Female Genital Mutilation/vaginal surgery which is unreversed (assessed antenatally)
* Women with clotting disorders; either longstanding or following intrapartum events
* Women who have just had, or are having an ongoing PPH
* Women in whom the third stage of labour is not complete (placenta remains in situ).
* Women who have had a caesarean section

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants for whom the PPH Butterfly is the correct size | Up to 8 weeks
  This outcome measure will be assessed through the use of a Likert scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Weeks, Principal Investigator — University of Liverpool
Locations (1):
- Liverpool Womens Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No